CLINICAL TRIAL: NCT06919900
Title: Motor Learning of Fall Resistant Skills Through Slip and Trip Exposure in Multiple Sclerosis
Acronym: STRES-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Feng Yang, PhD, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H25443
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (Relapsing Remitting)
Keywords: Falls; Fall prevention; Slips; Trips
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participants and outcome assessors will be blinded to each participant's group assignment. However, the researchers who conduct the training will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): During the acquisition session, this group will undergo perturbation training on the treadmill while wearing a safety harness. Then, they will experience an unexpected slip and trip while wearing a safety harness and walking overground. During the 3-month and 6-month retention sessions, they will experience a slip and trip during treadmill walking and a slip and trip during overground walking.
  Interventions: Behavioral: Perturbation Training
- Control Group (Active Comparator): During the acquisition session, this group will walk on the treadmill without perturbations for the same amount of time as the training group. Then, they will experience an unexpected slip and trip while wearing a safety harness and walking overground. During the 3-month and 6-month retention sessions, they will experience a slip and trip during treadmill walking and a slip and trip during overground walking.
  Interventions: Behavioral: Treadmill Walking

INTERVENTIONS:
Behavioral: Perturbation Training — Unexpected slips blended with trips and unperturbed walking trials on a treadmill. A safety harness will be worn at all times.
  Arms: Training Group
Behavioral: Treadmill Walking — Treadmill walking for the same amount of time as the training group without perturbation. A safety harness will be worn at all times.
  Arms: Control Group

SUMMARY:
The primary purpose of this interventional study is to examine the overall motor learning capacity from exposure to repeated perturbations among ambulatory people with multiple sclerosis (MS). This project will advance our understanding of learning new motor skills from exposure to external perturbations. If it is proven that people with MS can learn motor skills from perturbation training, the findings from this study will pave a theoretical foundation for applying perturbation training as a promising fall prevention intervention for people with MS.

DETAILED DESCRIPTION:
Falls present a significant health risk for people with multiple sclerosis (PwMS). Perturbation training has emerged as a promising strategy to prevent falls. This type of training, which is based on sensorimotor adaptation and motor learning, capitalizes on the central nervous system's (CNS) ability to develop new motor skills. With repeated exposure to large-scale slip or trip perturbations, participants can quickly learn how to better respond to falls. The primary benefits of this training include improved dynamic stability control, both proactively and reactively, by adjusting the body's center of mass (COM) relative to its base of support (BOS).

Sixty-four individuals with relapsing-remitting multiple sclerosis (MS) will be randomly assigned to one of two groups: Group A (training) and Group B (control). Both groups will first participate in an acquisition session. Group A will undergo a training procedure blending slips, trips, and unperturbed walking on a treadmill. In contrast, Group B will walk on the treadmill for the same duration without any perturbations. Immediately following the acquisition session, both groups will experience an unexpected slip and trip while walking over ground (with the order of the slip and trip randomized). Three and six months later, both groups will complete two retention sessions. Each retention session will involve experiencing a treadmill slip and trip (treadmill reslip and retrip) and an overground slip and trip (overground reslip and retrip), with the order randomized. Responses to these perturbations will be measured using the outcomes of fall or non-fall, dynamic stability, leg muscle reaction times, and recovery step length. Additionally, real-life prospective falls and near falls will be monitored for both groups over the six months following the acquisition session.

This project will advance our understanding of learning new motor skills from exposure to external perturbations. If it is proven that people with MS can learn motor skills from perturbation training, the findings from this study will pave a theoretical foundation for applying perturbation training as a promising fall prevention intervention for people with MS.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed multiple sclerosis
2. At least 45 years old
3. Able to walk independently at least 25 feet
4. Able to stand independently for at least 30 seconds
5. Patient Determined Disability Steps score between 0 and 4
6. Free from pregnancy
7. Montreal Cognitive Assessment score of 23 or higher

Exclusion Criteria:

1. Previous experience with perturbation training
2. T-score from the dual x-ray absorptiometry (DXA) scan of less than -2.5
3. Coexisting psychiatric disorders or other neurological conditions, severe medical illness, or cardiovascular diseases
4. Participants have had a relapse in the past 8 weeks

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Perturbation Outcome (Fall or Non-Fall) on the Treadmill or Overground | Baseline (acquisition session), 3-month retention session, 6-month retention session.
  A loadcell will be connected to the safety harness (above the participant's head) and will measure the force exerted on the safety harness during each perturbation trial. Perturbation outcomes will be classified as falls if the peak loadcell force exceeds 30% of the body weight. Otherwise, perturbation outcomes will be classified as non-falls.

SECONDARY OUTCOMES:
Dynamic Gait Stability as defined by the Feasible Stability Region (FSR) Theory | Baseline (acquisition session), 3-month retention session, 6-month retention session.
  FSR-based dynamic gait stability considers both the center of mass position and velocity during the slip or trip recovery process. Dynamic stability will be calculated at the foot touchdown before and after the perturbation onset. For slip-falls (or trip-falls), the larger (or smaller) the stability value, the more stable one is in resisting slip-related backward (or trip-induced forward) falling.
Leg Muscle Reaction Time | Baseline (acquisition session), 3-month retention session, 6-month retention session.
  The reaction times will be determined as the duration from the perturbation onset to the instant when the respective muscle is activated.
Recovery Step Length | Baseline (acquisition session), 3-month retention session, 6-month retention session.
  Recovery step length will be calculated as the distance between the heels at recovery foot touchdown and normalized to body height.
Prospective Real-Life Falls and Near Falls | 6 month period after the acquisition session
  Both groups will report their fall or near-fall incidents through an online survey weekly.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia State University Biomechanics Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang F, Pai YC. Automatic recognition of falls in gait-slip training: Harness load cell based criteria. J Biomech. 2011 Aug 11;44(12):2243-9. doi: 10.1016/j.jbiomech.2011.05.039. Epub 2011 Jun 21. PMID 21696744
- [Background] Yang F, Bhatt T, Pai YC. Generalization of treadmill-slip training to prevent a fall following a sudden (novel) slip in over-ground walking. J Biomech. 2013 Jan 4;46(1):63-9. doi: 10.1016/j.jbiomech.2012.10.002. Epub 2012 Nov 8. PMID 23141636
- [Background] Yang F, Su X, Wen PS, Lazarus J. Adaptation to repeated gait-slip perturbations among individuals with multiple sclerosis. Mult Scler Relat Disord. 2019 Oct;35:135-141. doi: 10.1016/j.msard.2019.07.019. Epub 2019 Jul 23. PMID 31376685